CLINICAL TRIAL: NCT03283280
Title: Clinical Performance of Short Fiber Reinforced Resin Composite Restorations Versus Indirect Nanohybrid Resin Composite Onlay Restorations in Complex Proximal Cavities of Molars
Brief Title: Clinical Performance of Short Fiber Reinforced Resin Composite Versus Indirect Nanohybrid Resin Composite Onlay Restorations.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawda Hesham Abd ElAziz, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-10-9-2017
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: Short fiber reinforced resin composite; Nanohybrid resin composite; Indirect resin composite restoration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be blinded to the material type
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short fiber RC (Experimental): Short fiber reinforced resin composite restoration (Ever X Posterior, Gc Europe) that is used in high stress bearing areas as direct onlay restoration.
  Interventions: Other: Ever X Posterior
- Nanohybrid RC (Active Comparator): Nanohybrid resin composite (GrandioSO, VOCO GmbH Germany ) that can be used to make indirect restorations in posterior teeth.
  Interventions: Other: Ever X Posterior

INTERVENTIONS:
Other: Ever X Posterior — Resin composite restoration can be made as a direct onlay
  Other Names: Short fiber reinforced resin composite

SUMMARY:
clinical performance of short fiber reinforced resin composite versus indirect nanohybrid resin composite onlay restorations in complex proximal cavities of molar teeth will be evaluated over one year.

DETAILED DESCRIPTION:
Resin composite materials have been rapidly developed in the latest few years. Direct resin composite restorations become the golden standard for restoring intracoronal cavities. While for the extracoronal cavities, the indirect resin composite onlays tend to replace metallic restorations in most situations being more esthetic and conservative with lower cost (Rocca & Krejci, 2007).

Indirect resin composite onlays usually are lab processed in two appointments but it can be made in one appointment through CAD/CAM technology or by flexible model technique (semidirect technique).

These restorations offer more control on the proximal contacts and the anatomic form over the direct approach. Polymerization shrinkage occurs outside the patient mouth so the stresses are decreased and become limited to the width of the luting space. Annual failure rate (AFR) of indirect posterior resin composite restorations is up to 10% (Manhart et al, 2004).

One of the advancement in resin composite technology is the evolution of short fiber reinforced resin composite (SFRC) material that allows making a direct onlay restoration possible thus offers less procedural steps and saves more time (Garoushi et al, 2013).

This material is made to be used as a dentine substitute in the high stress-bearing areas. It is covered by a conventional resin composite filling to act as the enamel replacement this combination gives us a kind of biomimetic restoration.

ELIGIBILITY:
Inclusion Criteria

1. Pulp asymptomatic vital carious upper or lower molars.
2. Proximal complex carious cavities involving one or two weak cusps.
3. Replacement of old amalgam or resin composite restoration due to recurrent caries or either tooth or restoration fracture.
4. Presence of favorable occlusion.
5. Healthy volunteers

Exclusion Criteria:

1. Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.
2. Deep subgingival cavity margins.
3. Possible future prosthodontic restoration of teeth.
4. Severe periodontal problems.
5. Medically compromised patients.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in the Clinical performance | Change from the Baseline at six months and 12 months.
  Measured using modified USPHS criteria for clinical evaluation of restoration failure

CONTACTS AND LOCATIONS:
Overall Officials: Rawda Hesham Abd ElAziz, Msc, Principal Investigator — Assistant lecturer
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Short fiber reinforced resin composite — http://www.gceurope.com/products/everxposterior/
- See also: Indirect nanohybrid resin composite — http://www.voco.com/us/product/GrandioSO/index.html